CLINICAL TRIAL: NCT03126201
Title: Predictors of Disease Progression in Patients With Primary Focal Segmental Glomerulosclerosis
Brief Title: Predictors of Disease Progression in Primary Focal Segmental Glomerulosclerosis
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Associate Professor of Medicine, Istanbul University
Other Study IDs: 333
Record Dates: First submitted 2017-04-16; First posted 2017-04-24 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Glomerulonephritis; Focal Segmental Glomerulosclerosis
Keywords: focal segmental glomerulosclerosis; disease progression
MeSH Terms: conditions — Glomerulonephritis; Glomerulosclerosis, Focal Segmental; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with biopsy-proven primary focal segmental glomerulosclerosis.

SUMMARY:
Focal segmental glomerulosclerosis (FSGS) is one of the most common primary glomerular diseases leading to end stage renal disease. In this study, our aim is to evaluate the effects of histopathological, clinical, and laboratory features of patients with primary FSGS on the disease progression.

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) is one of the most common primary glomerular diseases leading to end stage renal disease worldwide. Numerous studies have been conducted in order to identify the etiology of this debilitating disease. Beyond the etiological research, however, few studies managed to demonstrate the possible predictors of disease progression in patients. Therefore, we aim to evaluate the effects of histopathological, clinical, and laboratory features of patients with primary FSGS on the disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven primary focal segmental glomerulosclerosis.
* Patients who have a renal biopsy available for reviewing including 8 or more glomeruli.
* Patients who have been followed-up for at least 6 months or have progressed to primary outcome regardless the duration of follow-up.

Exclusion Criteria:

* Patients who have secondary focal segmental glomerulosclerosis attributable to any other condition (e.g., obesity, HIV, relevant drug exposure).
* Patients who have a genetic mutation or variation creating a tendency for developing focal segmental glomerulosclerosis.
* Patients who are unwilling or unable to consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven primary focal segmental glomerulosclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Reduction in kidney function and/or progression to end stage renal disease | 5-10 years
  At least a fifty-percent reduction in baseline estimated glomerular filtration rate (eGFR) or development of kidney failure, which was defined as a category G5 CKD (eGFR <15 ml/min/1.73 m2).

SECONDARY OUTCOMES:
Complete remission | 5-10 years
  Proteinuria below 0.5 g/24h and an eGFR of ≥60 ml/min per 1.73 m2 (or a return of ±15% of baseline values in those with eGFR <60 ml/min per 1.73 m2).
Partial remission | 5-10 years
  Absence of complete remission, proteinuria reduction of >50% (and a proteinuria value of <3 g/24h in patients with nephrotic range proteinuria at baseline), and stabilization (±25%) or improvement in renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Agati VD, Kaskel FJ, Falk RJ. Focal segmental glomerulosclerosis. N Engl J Med. 2011 Dec 22;365(25):2398-411. doi: 10.1056/NEJMra1106556. No abstract available. PMID 22187987